CLINICAL TRIAL: NCT04325100
Title: Development and Validation of an Intervention Targeting Motivational Negative Symptoms: Switch Protocol 2
Brief Title: Intervention Targeting Motivational Negative Symptoms
Acronym: Switch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Principal Investigator, Thonon Bénédicte, Principal investigator, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B707201629105
Record Dates: First submitted 2020-03-19; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Masking Description: A blinding procedure was used for the evaluation of the Brief Negative Symptom Scale: interviews were recorded and each video or sound recording was evaluated at the end of the study by one (or two) independent evaluator who was unaware of the recordings' assessment time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switch - i (Experimental): Individual sessions
  Interventions: Behavioral: Switch - Individual sessions
- Switch - g (Experimental): Group programme
  Interventions: Behavioral: Switch - Group programme

INTERVENTIONS:
Behavioral: Switch - Individual sessions — Participants follow the Switch intervention through individual sessions (1 hour, twice a week, for around 2 months).
  Participants are provided with a folder which presents the rational for each strategy. Take-home assignments are given and stored in the same folder. Participants are also given small cards (that can fit in their wallet) containing the key elements of each strategy.
  The intervention manual can be obtained from the main investigator (in French).
  Arms: Switch - i
Behavioral: Switch - Group programme — Participants follow the Switch group programme (2 hours, twice a week, for around 2 months).
  During the group sessions, a powerpoint presentation and different media are used to present the different parts of the motivation model. Participants learn the different strategies (e.g., cognitive defusion, pleasure anticipation, problem solving) through individual and group exercises.
  Participants are provided with a folder which presents the rational for each strategy. Take-home assignments are given and stored in the same folder. Participants are also given small cards (that can fit in their wallet) containing the key elements of each strategy.
  The intervention manual and the presentation material can be obtained from the main investigator (in French).
  Arms: Switch - g

SUMMARY:
This study aims to investigate the effects of the Switch intervention on motivation and associated processes and explore the dynamics between the processes.

A single case approach is followed, with a pre-post and follow-up assessment design, and continuous ambulatory assessments (experience sampling method (ESM) and step count).

DETAILED DESCRIPTION:
Motivational negative symptoms hinder quality of life and daily functioning of individuals with schizophrenia spectrum, bipolar and major depressive disorders.

A recently developed intervention, Switch, has shown promising effects on negative symptoms and functional outcomes. Switch is based on a model that identifies various cognitive, behavioural and emotional processes related to motivation and goal-directed behaviours: pleasure anticipation, value-effort-probability computation, (dys)functional attitudes (e.g., discouraging thoughts, self-efficacy), planning, initiation, in-the-moment enjoyment, reminiscence. The intervention combines a person-centred and recovery approach with cognitive, behavioural and 3rd wave techniques to tackle the obstacles related to motivation and goal-directed behaviours (i.e., targetting the various cognitive, behavioural and emotional processes listed above). Thus, an important part of the intervention focuses on the person's strengths, needs, goals and values. Furthermore, various strategies (e.g., cognitive defusion, pleasure anticipation, problem solving, reminiscence) are used to encourage engagement in meaningful personal goals and values.

The Switch intervention is provided either in individual (one-hour sessions), or in a group setting (two-hour sessions), twice a week for around two months.

There are three types of evaluation: traditional assessment scales of motivational deficits, apathy, quality of life and daily functioning (pre, post and follow-up at 3 months); ambulatory assessment including ESM (i.e., daily questionnaires); actigraphy (step count).

The aims of this study is to evaluate the efficacy of Switch in two different settings (i.e., individual sessions and a group programme) on motivation/apathy and functional outcomes/quality of life. Furthermore, we wish to explore the effects of Switch on process related to motivation and goal-directed behaviours (e.g., pleasure anticipation, reminiscence, defeatist beliefs, activities' meaningfulness) and on activity (i.e., step count). Finally, we wish to evaluate the dynamics between the different cognitive, behavioural and emotional processes related to motivation and goal-directed behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-V (DSM-V) criteria for schizophrenia, schizoaffective, bipolar or major depressive disorder (American Psychiatric Association, 2013).
* Good understanding of French.

Exclusion Criteria:

* Presenting an unstable clinical picture;
* Evidence of a significant change in medication within one month prior to baseline assessment;
* Having a history of severe brain trauma or epilepsy;
* Comorbid intellectual disability;
* Moderate or severe substance use disorder other than tobacco (according to the DSM-V; i.e., showing 4 or more symptoms).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Brief Negative Symptom Scale (BNSS) | Baseline
  There are 13 items that are scored from 0 to 6 (0 = no impairment; 1 = very slight; 2 = mild; 3 = moderate; 4 = moderately severe; 5 = marked; 6 = severe). The Expressive deficit factor includes the following subscales: Blunted affect (facial expression, vocal expression, expressive gestures) and Alogia (quantity of speech, spontaneous elaboration).Each item is scored from 0 to 6 (0 = no impairment; 1 = very slight; 2 = mild; 3 = moderate; 4 = moderately severe; 5 = marked; 6 = severe).
Brief Negative Symptom Scale (BNSS) | 2 months (post intervention)
  There are 13 items that are scored from 0 to 6 (0 = no impairment; 1 = very slight; 2 = mild; 3 = moderate; 4 = moderately severe; 5 = marked; 6 = severe). The Expressive deficit factor includes the following subscales: Blunted affect (facial expression, vocal expression, expressive gestures) and Alogia (quantity of speech, spontaneous elaboration).Each item is scored from 0 to 6 (0 = no impairment; 1 = very slight; 2 = mild; 3 = moderate; 4 = moderately severe; 5 = marked; 6 = severe).
Brief Negative Symptom Scale (BNSS) | 6 months (follow-up)
  There are 13 items that are scored from 0 to 6 (0 = no impairment; 1 = very slight; 2 = mild; 3 = moderate; 4 = moderately severe; 5 = marked; 6 = severe). The Expressive deficit factor includes the following subscales: Blunted affect (facial expression, vocal expression, expressive gestures) and Alogia (quantity of speech, spontaneous elaboration).Each item is scored from 0 to 6 (0 = no impairment; 1 = very slight; 2 = mild; 3 = moderate; 4 = moderately severe; 5 = marked; 6 = severe).
Lille Apathy Rating Scale (patient version) (LARS-p) | Baseline
  The LARS is a semi-structured interview designed to evaluate the different dimensions (cognitive, emotional and behavioural) of apathy in schizophrenia, through the following subscales: Everyday productivity, Interests, Taking initiatives, Novelty seeking, Voluntary actions, Emotional responses, Concern, Social life and Self-awareness. The total score ranges from -36 to 36 ([-36; -22] = absence of apathy; [-21; -17] = tendency towards apathy; [-16; -10] = moderate apathy; [-9; 36] = severe apathy).
Lille Apathy Rating Scale (patient version) (LARS-p) | 2 months (post-intervention)
  The LARS is a semi-structured interview designed to evaluate the different dimensions (cognitive, emotional and behavioural) of apathy in schizophrenia, through the following subscales: Everyday productivity, Interests, Taking initiatives, Novelty seeking, Voluntary actions, Emotional responses, Concern, Social life and Self-awareness. The total score ranges from -36 to 36 ([-36; -22] = absence of apathy; [-21; -17] = tendency towards apathy; [-16; -10] = moderate apathy; [-9; 36] = severe apathy).
Lille Apathy Rating Scale (informant version) (LARS-i) | 6 months (follow-up)
  The LARS is a semi-structured interview designed to evaluate the different dimensions (cognitive, emotional and behavioural) of apathy in schizophrenia, through the following subscales: Everyday productivity, Interests, Taking initiatives, Novelty seeking, Voluntary actions, Emotional responses, Concern, Social life and Self-awareness. The total score ranges from -36 to 36 ([-36; -22] = absence of apathy; [-21; -17] = tendency towards apathy; [-16; -10] = moderate apathy; [-9; 36] = severe apathy).
Schizophrenia - Quality of Life questionnaire | Baseline (month 0)
  The S-QoL is a 41-item questionnaire that evaluates life satisfaction regarding psychological wellbeing, self-esteem, family relationships, relationships with friends, resilience, physical wellbeing, autonomy and sentimental life. Items are rated on a 5-point Likert scale (1 = much less satisfied than expected; 2 = less satisfied; 3 = slightly less satisfied; 4 = as satisfied; 5 = more satisfied). The total score ranges from 0 to 100, higher scores indicating better subjective quality of life.
Schizophrenia - Quality of Life questionnaire | 2 months (post-intervention)
  The S-QoL is a 41-item questionnaire that evaluates life satisfaction regarding psychological wellbeing, self-esteem, family relationships, relationships with friends, resilience, physical wellbeing, autonomy and sentimental life. Items are rated on a 5-point Likert scale (1 = much less satisfied than expected; 2 = less satisfied; 3 = slightly less satisfied; 4 = as satisfied; 5 = more satisfied). The total score ranges from 0 to 100, higher scores indicating better subjective quality of life.
Schizophrenia - Quality of Life questionnaire | 6 months (follow-up)
  The S-QoL is a 41-item questionnaire that evaluates life satisfaction regarding psychological wellbeing, self-esteem, family relationships, relationships with friends, resilience, physical wellbeing, autonomy and sentimental life. Items are rated on a 5-point Likert scale (1 = much less satisfied than expected; 2 = less satisfied; 3 = slightly less satisfied; 4 = as satisfied; 5 = more satisfied). The total score ranges from 0 to 100, higher scores indicating better subjective quality of life.
Functional Remission of General Schizophrenia (FROGS) | Baseline
  The FROGS is a measure of daily life outcomes, which evaluates level of functioning in 5 different domains: Daily life, Activities, Relationships, Quality of adaptation, and Health and treatment. The total score ranges from 19 to 95. The threshold score for remission is 61.
Functional Remission of General Schizophrenia (FROGS) | 2 months (post-intervention)
  The FROGS is a measure of daily life outcomes, which evaluates level of functioning in 5 different domains: Daily life, Activities, Relationships, Quality of adaptation, and Health and treatment. The total score ranges from 19 to 95. The threshold score for remission is 61.
Functional Remission of General Schizophrenia (FROGS) | 6 months (follow-up)
  The FROGS is a measure of daily life outcomes, which evaluates level of functioning in 5 different domains: Daily life, Activities, Relationships, Quality of adaptation, and Health and treatment. The total score ranges from 19 to 95. The threshold score for remission is 61.

SECONDARY OUTCOMES:
Experience Sampling Method | Baseline (14 days): 5 triggers/day
  Questionnaire including 14 questions regarding mood, discouraging beliefs, coping, confidence, motivation, energy, social environment, current activity, initiation, present enjoyment, activity's meaning, effort, reminiscence, projection into the future. The questionnaires are sent 3 times (intervention phase) or 5 times per day (baseline, post-intervention and follow-up phases).
Experience Sampling Method | Intervention phase (60 days): 3 triggers/day
  Questionnaire including 14 questions regarding mood, discouraging beliefs, coping, confidence, motivation, energy, social environment, current activity, initiation, present enjoyment, activity's meaning, effort, reminiscence, projection into the future. The questionnaires are sent 3 times (intervention phase) or 5 times per day (baseline, post-intervention and follow-up phases).
Experience Sampling Method | Post-intervention (14 days): 5 triggers/day
  Questionnaire including 14 questions regarding mood, discouraging beliefs, coping, confidence, motivation, energy, social environment, current activity, initiation, present enjoyment, activity's meaning, effort, reminiscence, projection into the future. The questionnaires are sent 3 times (intervention phase) or 5 times per day (baseline, post-intervention and follow-up phases).
Experience Sampling Method | Follow-up (14 days): 5 triggers/day
  Questionnaire including 14 questions regarding mood, discouraging beliefs, coping, confidence, motivation, energy, social environment, current activity, initiation, present enjoyment, activity's meaning, effort, reminiscence, projection into the future. The questionnaires are sent 3 times (intervention phase) or 5 times per day (baseline, post-intervention and follow-up phases).
Step count | Baseline (14 days): 5 triggers/day
  Daily step count (total per day) via an activity band.
Step count | Intervention phase (60 days): 3 triggers/day
  Daily step count (total per day) via an activity band.
Step count | Post-intervention (14 days): 5 triggers/day
  Daily step count (total per day) via an activity band.
Step count | Follow-up (14 days): 5 triggers/day
  Daily step count (total per day) via an activity band.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Laroi, PhD, Study Director — University of Liege
Locations (1):
- University of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data and analyses will be available from an online repository or from the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Thonon B, Van Aubel E, Lafit G, Della Libera C, Laroi F. Idiographic analyses of motivation and related processes in participants with schizophrenia following a therapeutic intervention for negative symptoms. BMC Psychiatry. 2020 Sep 25;20(1):464. doi: 10.1186/s12888-020-02824-5. PMID 32977798